CLINICAL TRIAL: NCT01598584
Title: A Phase II/III Prospective Randomized Placebo-control Trail Compare Mirtazapine Plus Gemcitabine With Gemcitabine in Metastasis Pancreatic Cancer
Brief Title: Mirtazapine Plus Gemcitabine Versus Gemcitabine in Metastasis Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Gemcitabine is not the first choice for most pancreatic cancer patients nowdays
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TJ20111123
Record Dates: First submitted 2012-05-05; First posted 2012-05-15 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2012-12

CONDITIONS: Pancreatic Cancer
Keywords: Mirtazapine; gemcitabine; placebo; RCT; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Mirtazapine; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo plus gemcitabine (Placebo Comparator): we design placebo plus gemcitabine as control arm
  Interventions: Drug: Gemcitabine, placebo
- Mirtazapine plus gemcitabine (Experimental): We design Mirtazapine plus gemcitabine as experimental arm
  Interventions: Drug: Mirtazapine plus gemcitabine

INTERVENTIONS:
Drug: Mirtazapine plus gemcitabine — Mirtazapine,15mg/day for 3 days, If patients is durable, the dosage increase to 30mg/day, if the patient is durable, the doctor then will decided whether to increase to 45mg. Gemcitabine 1000mg/M2,d1,d8,q3w
  Other Names: Mirtazapine; Gemcitabine; pancreatic cancer
  Arms: Mirtazapine plus gemcitabine
Drug: Gemcitabine, placebo — Gemcitabine 1.0g/m2,d1,d8,q3w placebo
  Other Names: placebo; Gemcitabine; pancreatic cancer; randomised control trial
  Arms: placebo plus gemcitabine

SUMMARY:
Depression and anxiety accompany with advanced cancer. The effect of anti-anxiety depression has not evaluated in special cancers. Mirtazapine is a drug anti-anxiety depression and has a high risk increase weight. So the investigators assume Mirtazapine would not only improve the anxiety and depression of metastasis pancreas cancer but also would improve the appetite of such patients which would improve dyscrasia of pancreas cancer patients. The drug may improve the quality of life in advanced pancreatic cancer which is of short survival.

DETAILED DESCRIPTION:
The investigators design a phase II/III trial to compared Mirtazapine plus gemcitabine with gemcitabine in metastasis pancreatic cancer. The investigators planed to enroll 33 patients for each arm after randomization.

The inclusion criteria included:

1. Patients shall have normal organic function such as liver function, Cardiac function and renal function.
2. Before enrolled, anxious and depression states will be evaluated by the Hamilton degree of depression and anxiety scale. Only patients with definite depression and/or anxiety will be considering participating this trial.
3. Pancreatic cancer patients with ECOG 1～2 scores will be enrolled.
4. Patients should be expected to live no shorter than 1.5 months

The investigators will evaluated the quality of life by SF-36 scale as primary outcome. The second outcomes include anxious and depression scores, objective response rate, progress free survival, overall Survival and chemotherapy induced nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of pancreatic cancer shall have normal organic function such as liver function, cardiac function and renal function.
2. Before enrolled, anxious and depression states will be evaluated by the Hamilton degree of depression and anxiety scale. Only patients with definite depression and/or anxiety will be considering participating this trial.
3. Pancreatic cancer patients with ECOG 1～2 scores will be enrolled.
4. Patients should be expected to live no shorter than 1.5 months

Exclusion Criteria:

1. Patients receiving other anti-cancer drugs;
2. Patients who discontinue anti-cancer drugs less than 4 weeks, for patients who received Postoperative adjuvant chemotherapy less than 6 weeks. Shorter than 4 weeks after operation;
3. Patient with inadequate Blood system,liver function and renal function.
4. Brain metastasis is of symptoms
5. Patient with arrhythmia,myocardial ischemia,serious atrioventricular block,inadequate cardiac function,serious valvular heart disease;
6. Chronic enteritis or intestinal obstruction
7. Bone marrow failure
8. Mental disease difficult to control
9. Participated other clinic trial within 3 months
10. Pregnant or lactation patients
11. The researcher evaluate the patient is not suitable for this trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
quality of life | up to 3 years
  primary outcome is the quality of life evaluated by SF-36 scale

SECONDARY OUTCOMES:
anxiety and depression scores | up to 3 years
  The second outcomes include anxious and depression scores
objective response rate | up to 3 years
progress free survival, | up to 3 years
overall Survival | up to 3 years
chemotherapy induced nausea and vomiting | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, MD, PHD, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- TianjinCIH, Tianjin, Tianjin Municipality, China